CLINICAL TRIAL: NCT02125630
Title: The Effect of Primary Surgery in Patients With Stage IV Breast Cancer With Bone Metastasis Only
Brief Title: Bone Metastasis and Surgery in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Federation of Breast Diseases Societies (Other)
Responsible Party: Sponsor
Other Study IDs: BOMET MF14-01; PROTOCOL BOMET MF14-01 (Other: TURKISH FEDERATION OF BREAST DISEASE SOCITIES)
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Surgery
Keywords: Metastatic breast carcer; Bone metastasis; surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative; Mastectomy; Mastectomy, Segmental; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Systemic therapy: Standart chemotherapy
  Interventions: Drug: Systemic therapy
- Primary surgery: Standart surgery
  Interventions: Procedure: Surgery
- Neoadjuvant chemotherapy: Standart chemotherapy followed by surgery
  Interventions: Procedure: Surgery; Drug: Systemic therapy

INTERVENTIONS:
Procedure: Surgery — Surgery to primary tumor
  Other Names: mastectomy, lumpectomy
  Groups: Neoadjuvant chemotherapy; Primary surgery
Drug: Systemic therapy — Systemic therapy based on tumor phenotype
  Other Names: Chemotherapy, hormone therapy, biphosphanetes
  Groups: Neoadjuvant chemotherapy; Systemic therapy

SUMMARY:
A registry trial evaluating resection of the primary breast tumor in women presenting with de novo stage IV breast cancer with bone metastasis only. Previous reports of carefully selected patients presenting with stage IV breast cancer suggest that surgery on the primary tumor may result in improved survival, but this remains unproven. The early results of our ongoing trial MF07-01 trial (a phase III randomized controlled trial of breast cancer women with distant metastases at presentation who receive loco-regional treatment for intact primary tumor compared with those who do not receive such treatment) showed that patients with bone metastasis only have a trend toward improved survival with initial surgery.

DETAILED DESCRIPTION:
This registry trial evaluating resection of the primary breast tumor in women presenting with de novo stage IV breast cancer with bone metastasis only. Previous reports of carefully selected patients presenting with stage IV breast cancer suggest that surgery on the primary tumor may result in improved survival, but this remains unproven. The early results of our ongoing trial MF07-01 trial (a phase III randomized controlled trial of breast cancer women with distant metastases at presentation who receive loco-regional treatment for intact primary tumor compared with those who do not receive such treatment) showed that patients with bone metastasis only have a trend toward improved survival with initial surgery. Our goal is to test if primary surgery improves overall survival in bone only metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast tumor amenable for complete surgical resection
* Patients in good physical condition for receiving protocol driven locoregional and systemic treatment
* Patients eligible for sentinel lymph node (SLN) biopsy and receiving radiotherapy.

Exclusion Criteria:

* Primary tumor not amenable for complete resection (such as tumor extending to neighboring tissues; T4a,c or inflammatory breast cancer; T4d)
* Primary tumor with extended infection, bleeding, or necrosis
* Patients with poor physical condition which prevents the patient from receiving protocol driven locoregional and systemic treatment
* Synchronous primary cancer at the contralateral breast
* Previous diagnosis of other cancers (excluding basal cell skin cancer
* Squamous cell skin cancer
* Cervical intraepithelial neoplasia)
* Clinically involved contralateral axillary nodes
* Patients not suitable for adequate follow-up
* Failure to give informed consent

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female patients diagnosed with de novo stage IV breast cancer
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Years

SECONDARY OUTCOMES:
Locoregional progression | 5 years
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Soran, MD, MPH, Study Chair — University of Pittsburgh; Serdar Ozbas, MD, Principal Investigator — Guven Hospital; Lutfi Doğan, MD, Principal Investigator — Ankara Onkoloji Hastanesi
Locations (1):
- Istanbul University Medical faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided